CLINICAL TRIAL: NCT00486759
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Trial Comparing the Efficacy of Bevacizumab in Combination With Rituximab and CHOP (R-CHOP + Bevacizumab) Versus Rituximab and CHOP (R-CHOP) in Previously Untreated Patients With CD20-positive Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: A Study of Bevacizumab (Avastin) in Combination With Rituximab (MabThera) and CHOP (Cyclophosphamide, Hydroxydaunorubicin [Doxorubicin], Oncovin [Vincristine], Prednisone) Chemotherapy in Patients With Diffuse Large B-cell Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to an unfavorable benefit/risk ratio.
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO20603
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Bevacizumab; Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Bevacizumab + rituximab + CHOP (Experimental): Patients received bevacizumab 5 mg/kg/week on Day 1 of each cycle + rituximab 375 mg/m^2 intravenously (IV) on Day 1 of each cycle + CHOP (cyclophosphamide, hydroxydaunorubicin [doxorubicin], Oncovin [vincristine], prednisone).
  Interventions: Drug: Bevacizumab; Drug: Rituximab; Drug: CHOP
- Placebo + rituximab + CHOP (Active Comparator): Patients received placebo to bevacizumab on Day 1 of each cycle + rituximab 375 mg/m^2 intravenously (IV) on Day 1 of each cycle + CHOP (cyclophosphamide, hydroxydaunorubicin [doxorubicin], Oncovin [vincristine], prednisone).
  Interventions: Drug: Rituximab; Drug: CHOP; Drug: Placebo

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab was administered at a dose of 15 mg/kg IV on Day 1 of each 21-day cycle for 8 cycles or at a dose 10 mg/kg IV on Day 1 of each 14-day cycle for 8 cycles. The cycle duration (14- or 21-day) was chosen by each center prior to initiation of the study and was the same for all patients enrolled at that center.
  Other Names: Avastin
  Arms: Bevacizumab + rituximab + CHOP
Drug: Rituximab — Rituximab was administered at a dose of 375 mg/m^2 IV on Day 1 of each 14- or 21-day cycle for 8 cycles. The cycle duration (14- or 21-day) was chosen by each center prior to initiation of the study and was the same for all patients enrolled at that center.
  Other Names: MabThera
Drug: CHOP — Cyclophosphamide was administered at a dose of 750 mg/m^2 IV on Day 1 of each cycle. Doxorubicin was administered at a dose of 50 mg/m^2 IV on Day 1 of each cycle. Vincristine was administered at a dose of 1.4 mg/m^2 IV (maximum of 2 mg) on Day 1 of each cycle. Prednisone was administered at a dose of 100 mg orally on Days 1-5 of each cycle. All 4 drugs were administered either every 21 days for 8 cycles or every 14 days for 6 cycles. The cycle duration (14- or 21-day) was chosen by each center prior to initiation of the study and was the same for all patients enrolled at that center.
Drug: Placebo — Placebo to bevacizumab was administered on Day 1 of each 14- or 21-day cycle for 8 cycles. The cycle duration (14- or 21-day) was chosen by each center prior to initiation of the study and was the same for all patients enrolled at that center.
  Arms: Placebo + rituximab + CHOP

SUMMARY:
This 2-arm study was designed to compare the efficacy and safety of bevacizumab (Avastin) in combination with rituximab (MabThera) and CHOP (cyclophosphamide, hydroxydaunorubicin [doxorubicin], Oncovin [vincristine], prednisone) chemotherapy (R-CHOP) versus rituximab plus CHOP chemotherapy (R-CHOP) in previously untreated patients with CD20-positive diffuse large B-cell lymphoma (DLBCL). Patients were randomized to receive 8 cycles of treatment with R-CHOP plus bevacizumab or R-CHOP plus placebo. Treatment with bevacizumab/placebo and R-CHOP was given either on a 2-week or 3-week schedule and bevacizumab was given at a weekly average dose of 5 mg/kg (10 mg/kg for 2-week cycles and 15 mg/kg for 3-week cycles).

DETAILED DESCRIPTION:
An independent Data and Safety Monitoring Board (DSMB) was established to review safety data collected during the study on an ongoing basis. At its meeting in December 2009, the DSMB noted a trend for increased cardiac toxicity in the experimental arm (R-CHOP + bevacizumab) compared with the control arm (R-CHOP + placebo). Additional efficacy analyses of data from 720 randomized patients were presented at a DSMB meeting on May 22, 2010; they indicated no improvement in efficacy with the addition of bevacizumab to R-CHOP. It was noted, however, that there was an apparent increase in the risk of cardiotoxicity, premature treatment withdrawal, serious adverse events (SAEs), fatal adverse events (AEs), and perforation/ulcer in the experimental arm. Based on its assessment of an increased risk with unlikely benefit for patients randomized to the experimental arm, the DSMB recommended that further enrollment in the study be permanently halted and that bevacizumab be discontinued for any patients randomized to the experimental arm. On May 31, 2010, the sponsor took the decision to stop enrollment into the study and the bevacizumab treatment was terminated with immediate effect as recommended by the DSMB.

The study protocol was amended. The primary objective of the study was changed from evaluation of efficacy to evaluation of safety and the study was extended to include an 18-month safety follow-up period. Because enrollment was terminated prematurely resulting in fewer enrolled patients than planned, the outcome measure data are premature due to fewer than expected events.

The time frame for the reporting of serious adverse events was modified. Serious adverse events (SAE) unrelated to study treatment were reported until 1 year post-treatment or until new anti-lymphoma treatment was initiated. SAEs judged to be related to study treatment and congestive heart failure events were reported at any time during the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ 18 and < 80 years of age.
* CD20-positive diffuse large B-cell lymphoma.
* Low-intermediate, high-intermediate, or high risk disease and/or bulky tumor (largest diameter ≥ 7.5 cm).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.

Exclusion Criteria:

* Prior treatment for diffuse large B-cell lymphoma.
* Types of non-Hodgkin's lymphoma other than diffuse large B-cell lymphoma (DLBCL).
* Central nervous system (CNS) involvement of lymphoma.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 787 (Actual)
Dates: Start 2007-07-26 (Actual); Primary Completion 2011-11-30 (Actual); Study Completion 2011-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (266):
- United States (17):
  - Uni of California - San Diego; Cancer Center & Dept of Medicine, La Jolla, California
  - Kenmar Research Inst., Whittier, California
  - University of Colorado Cancer Center Department of Hematology, Aurora, Colorado
  - Uni Medical Center; Division Of Hemotology/Oncology, Jacksonville, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - University of Kansas Medical Center; Department of Hematology, Kansas City, Kansas
  - St. Joseph Mercy Hospital; Department of Oncology, Ann Arbor, Michigan
  - Northeast Oncology Associates, Concord, North Carolina
  - Forsyth Regional Cancer Center; Piedmont Hematology/Oncology Associates, Winston-Salem, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - Charleston Cancer Center, Charleston, South Carolina
  - Uni of Texas Southwestern Medical Center, Dallas, Texas
  - Cancer Therapy & Research Center, San Antonio, Texas
  - Northwest Medical Specialties B, Federal Way, Washington
  - Rainier Physicians, Puyallup, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Argentina (4):
  - Hospital Italiano; Haemathology, Buenos Aires
  - Fundaleu; Haematology, Buenos Aires
  - Hospital Britanico; Haematology, Buenos Aires
  - HOSPITAL PRIVADO - CENTRO MEDICO DE CÓRDOBA; Dpto Oncología, Córdoba
- Australia (9):
  - Greenslopes Private Hospital; Gallipoli Research Centre, Greenslopes, Queensland
  - Princess Alexandra Hospital Woolloongabba; Clinical Hematology and Medical Oncology, Woolloongabba, Queensland
  - Royal Adelaide Hospital; Haematology, Institute of Medical Veterinary Science, Adelaide, South Australia
  - Ashford Cancer Center Research, Kurralta Park, South Australia
  - Frankston Hospital; Oncology/Haematology, Frankston, Victoria
  - Peter Maccallum Cancer Institute; Medical Oncology, Melbourne, Victoria
  - Alfred Hospital; Bone Marrow Transplant Unit, Melbourne, Victoria
  - Border Medical Oncology; Murray Valley Private Hospital, Wodonga, Victoria
  - Fremantle Hospital; Haematology, Fremantle, Western Australia
- Austria (3):
  - Lkh-Univ. Klinikum Graz; Klinik Für Innere Medizin I, Graz
  - Lkh Salzburg - Univ. Klinikum Salzburg; Iii. Medizinische Abt., Salzburg
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I - Hämatologie & Hämostaseologie, Vienna
- Brazil (8):
  - Centro Goiano de Oncologia - CGO, Goiânia, Goiás
  - Hospital de Caridade de Ijui; Oncologia, Ijuí, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS; Hematologia, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - UNICAMP, Campinas, São Paulo
  - Faculdade de Medicina do ABC - FMABC; Oncologia e Hematologia, Santo André, São Paulo
  - Santa Casa de Misericordia de Sao Paulo; Hematologia e Hemoterapia, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP; Hematologia, São Paulo, São Paulo
- Canada (18):
  - Tom Baker Cancer Centre; Dept of Medicine, Calgary, Alberta
  - Cross Cancer Institute ; Dept of Medical Oncology, Edmonton, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Health Science Centre, St. John's, Newfoundland and Labrador
  - QEII HSC; Oncology, Halifax, Nova Scotia
  - Cancer Centre of Southeastern Ontario; Kingston General Hospital, Kingston, Ontario
  - Credit Valley Hospital/Carlo Fidani Peel Regional Cancer Centre, Mississauga, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Hopital Charles Lemoyne; Centre Integre de Lutte Contre Le Cancer de La Monteregie, Greenfield Park, Quebec
  - Mcgill University - Royal Victoria Hospital; Oncology, Montreal, Quebec
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
  - Hopital de L'Enfant-Jesus; Hematology, Québec, Quebec
  - Chuq - Hopital Hotel Dieu de Quebec; Oncology, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre; Uni of Saskatoon Campus, Saskatoon, Saskatchewan
- China (12):
  - Cancer Hospital Chinese Academy of Medical Sciences., Beijing
  - Beijing Cancer Hospital, Beijing
  - Beijing Union Hospital, Beijing
  - General Hospital of Chinese PLA; Department of Hematology, Beijing
  - Fujian Cancer Hospital, Fuzhou
  - Fudan University Shanghai Cancer Center, Shanghai
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Changhai Hospital of Shanghai, Shanghai
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Institute of Hematology & Blood Diseases Hospital, Tianjin
  - The First Affiliated Hospital of The Fourth Military Medical University (Xijing Hospital), Xi'an
- Colombia (4):
  - Organizacion Sanitas Internacional, Bogotá
  - Hospital Pablo Tobon Uribe, Medellin-Antioquia
  - Instituto Cancerologia Medellin; Clinica Las Americas, Medellín
  - Oncólogos de Occidente, Pereira
- Czechia (6):
  - Fakultni nemocnice Brno; Interni hematoonkologicka klinika, Brno
  - Fn Hr. Kralove; IV. Interni Hematologicka Klinika, Hradec Králové
  - Fakultni nemocnice Olomouc; Hemato-onkologicka klinika, Olomouc
  - Fakultni Nemocnice Plzen, Hematologicko-Onkologicke Oddeleni, Plzen - Lochotin
  - Fakultní Nemocnice Královské Vinohrady; Hematologická Klinika, Prague
  - VshEOBECNÁ FAKULTNÍ NEMOCNICE; I. INTERNI KLINIKA, Prague
- Ecuador (3):
  - Teodoro Maldonado Carbo Hospital; Oncology Service, Guayaquil
  - Hospital Carlos Andrade Marin; Servicio de Oncología, Quito
  - Hospital Solca Quito; Oncologia, Quito
- France (33):
  - Clinique Claude Bernard; Onco Hematologie, Albi
  - Centre Hospitalier Uni Ire; Service de Medecine D, Angers
  - Institut Bergonie; Hematologie Oncologie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine; Chimiotherapie Radiotherapie, Bordeaux
  - Centre Francois Baclesse; Comite 2, Caen
  - Chu Estaing; Cons Hemato Medecine Interne, Clermont-Ferrand
  - Chu Site Du Bocage;Hematologie Clinique, Dijon
  - CH Dptal Les Oudairies; Hematologie Oncologie, La Roche-sur-Yon
  - Hopital Albert Michallon; Oncologie, La Tronche
  - Clinique Victor Hugo; Chimiotherapie, Le Mans
  - Hopital Claude Huriez; Hematologie, Lille
  - Hopital Uni Ire Dupuytren; Hematologie, Limoges
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Institut J Paolii Calmettes; Onco Hematologie 1, Marseille
  - Clinique Pont de Chaume; Oncologie Et Radiotherapie, Montauban
  - Hopital Saint Eloi; Hematologie Oncologie Medicale, Montpellier
  - Hopital de L'Archet; Hematologie Clinique, Nice
  - Polyclinique Kenval ; Radiotherapie Oncologie, Nîmes
  - Institut Curie; Oncologie Medicale, Paris
  - Hopital Saint Louis ; Service d Oncologie Medicale Fougere 6 (Pr Misset), Paris
  - Hopital Pitie Salpetriere; Hematologie Clinique, Paris
  - Hopital Saint Jean; Hematologie, Perpignan
  - Hopital De Haut Leveque; Hematologie Clinique, Pessac
  - Ch Lyon Sud; Hemato Secteur Jules Courmont, Pierre-Bénite
  - Hopital De La Miletrie; Hematologie Et Oncologie Medicale, Poitiers
  - Ch Jacques Puel;Oncologie Medicale, Rodez
  - ICL; Hematologie, Saint-Priest-en-Jarez
  - Hopital Sud; Hematologie Clinique, Salouël
  - Hopital Purpan; Hematologie Clinique, Toulouse
  - Clinique Pasteur; Oncologie Medicale, Toulouse
  - Hopital Bretonneau; Hematologie Therapie Cellulaire, Tours
  - Hopitaux De Brabois; Hematologie Medecine Interne, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy; Unite D'Hematologie, Villejuif
- Germany (43):
  - Gesundheitszentrum St. Marien GmbH; Med. II, Hämatologie/Onkologie, Amberg
  - Charité-Universitätsm. Berlin; Med. Klinik mit Schwerpunkt Hämatologie, Onkologie und Tumorimmunolo., Berlin
  - Charité; Onkologie & Hämatologie, Berlin
  - DIAKO Ev. Diakonie-Krankenhaus Bremen GmbH; Med. Klinik II; Hämatologie und internistische Onkologie, Bremen
  - Carl-Thiem-Klinik Cottbus; Medizinische Klinik, Cottbus
  - Klinikzentrum Mitte; Medizinische Klinik Gastroenterologie Haematologie / Onkologie, Dortmund
  - St. Johannes Hospital; Abt. Innere Medizin, Dortmund
  - St Antonius Hospital; Haematologie/Onkologie, Eschweiler
  - Krankenhaus Nordwest Medizinische Klinik, Frankfurt
  - Klinik Fulda; Abt. Itz, Fulda
  - Georg-August-Uniklinik ; Zentrum Innere Medizin Abt. Hämatologie & Onkologie, Göttingen
  - Universitätsklinikum Greifswald Klinik für Innere Medizin C und Poliklinik, Greifswald
  - Kath.Krankenhaus Hagen gem.GmbH St.-Marien-Hospital, Hagen
  - Asklepios Klinik St. Georg; Allgemeine Innere Medizin, Hamburg
  - Facharztzentrum Eppendorf, Studien GbR, Hamburg
  - Evang.Krankenhaus Abt. Hämatologie und Onkologie, Hamm
  - St.-Marien-Hospital Klinik Knappenstraße; Klinik für Hämatologie und Onkologie, Hamm
  - KRH Klinikum Siloah Medizinische Klinik III, Hanover
  - St. Bernward-Krankenhaus, Hildesheim
  - Universitaetsklinikum des Saarlandes; medizinische Klinik und Poliklinik; Innere Medizin I, Homburg/Saar
  - Städtisches Klinikum Karlsruhe gGmbH, II. Medizinische Klinik, Karlsruhe
  - St. Vincentius Kliniken Ag; Medizinische Klinik Abt. 2, Karlsruhe
  - Tagesklinik Landshut; Hämatologie/Onkologie, Landshut
  - Universitätsklinikum Leipzig Medizinische Klinik II Gastroenterolog. u. Hepatolog., Leipzig
  - Klinikum St.Georg gGmbH Klinik für Internistische Onkologie und Hämotologie, Leipzig
  - Klinikum der Stadt Ludwigshafen; Medizinische Klinik A, Ludwigshafen
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck, Med. Klinik I, Hämatologie/Onkologie, Lübeck
  - Märkische Kliniken GmbH, Klinikum Lüdenscheid; Hämatologie / Onkologie, Lüdenscheid
  - Otto von Guericke Uni Magdeburg Uniklinik; Hämatologie/Onkologie, Magdeburg
  - Klinikum Magdeburg gemeinnützige GmbH; Klinik Haematologie und Onkologie, Magdeburg
  - Klinikum Mannheim III. Medizinische Klinik, Mannheim
  - Klinikum der Universitaet Muenchen; Campus Großhadern; Medizinische Klinik III und Poliklinik, München
  - Westfälische Wilhelms-Universität Münster, Medizinische Klinik und Poliklinik A, Münster
  - Klinikum Oldenburg gGmbH; Klinik für Onkologie und Hämatologie, Oldenburg
  - Prosper-Hospital, Medizinische Klinik I, Recklinghausen
  - St Marien Krankenhaus; Medizinische Klinik Iii, Siegen
  - Klinikum Mutterhaus der Borromaeerinnen gGmbH; Haematologie/Onkologie, Trier
  - Krankenhaus der Barmherzigen Brüder Trier; Innere Medizin I, Hämatologie / Internistische Onkologie, Trier
  - Eberhard-Karls-Universität Tübingen; Medizinische Klinik I, Tübingen
  - Universitätsklinikum Ulm; Medizinische Uni-Klinik III Abt. Innere Medizin III Hämatologie u. Onkolo., Ulm
  - HSK Dr.-Horst-Schmidt-Kliniken; Innere Medizin I Kardiologie; Angiologie und Intensivmedizin, Wiesbaden
  - Helios Klinik Wuppertal; Medizinische Klinik I, Wuppertal
  - Kliniken St. Antonius; Zentrum Für Innere Medizin, Haematologie/Onkologie, Wuppertal
- Georgios Papanikolaou Hospital; Hematology Department, Thessaloniki, Greece
- Hong Kong (2):
  - Queen Elizabeth Hospital; Clinical Oncology, Hong Kong
  - Queen Mary Hospital; Dept of Medicine, Hong Kong
- Hungary (3):
  - Fov. Onk. Egyesitett Szent Istvan es Szent Laszlo Korhaz; Dept Of Bone Marrow Transplant, Budapest
  - National Institute of Oncology, A Dept of Internal Medicine, Budapest
  - University of Debrecen Medical and Health Science Center, Institute of Internal Medicine, Hematology, Debrecen
- Italy (15):
  - Irccs Ist. Tumori Giovanni Paolo Ii; Dipartimento Oncologia Medica, Bari, Apulia
  - A.O. Universitaria Policlinico S.Orsola-Malpighi Di Bologna, Bologna, Emilia-Romagna
  - Ospedale Regionale Di Parma; Divisione Di Oncologia Medica, Parma, Emilia-Romagna
  - Az. Osp. Arcispedale S. Maria Nuova; U.O. Di Ematologia, Reggio Emilia, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO); Dipartimento Di Oncologia Medica, Aviano, Friuli Venezia Giulia
  - A.O. Universitaria S. Maria Della Misericordia Di Udine; Oncologia; Clinica Ematologica, Udine, Friuli Venezia Giulia
  - Univ. Cattolica La Sapienza; Cattedra Di Ematologia, Rome, Lazio
  - ASST DI MONZA; Ematologia, Monza, Lombardy
  - Irccs Policlinico San Matteo; Divisione Di Ematologia, Pavia, Lombardy
  - Università Cattolica Del Sacro Cuore S.S. Giovanni Paolo Ii; Uoc Di Onco-Ematologia, Campobasso, Molise
  - Az. Osp. S. Luigi Gonzaga; Malattie Apparato Respiratorio 5 Ad Indirizzo Oncologico, Orbassano, Piedmont
  - A.O. Universitaria S. Giovanni Battista-Molinette Di Torino; Ematologia 1, Turin, Piedmont
  - Ospedale Ferrarotto; Divisione Di Ematologia, Via S. Sofia 78, Sicily
  - Ospedale Gen.Le Prov.Le 'C.G.Mazzoni'; Ematologia, Ascoli Piceno, The Marches
  - Ospedale Santa Chiara; Unita Operativa Di Ematologia, Pisa, Tuscany
- Lithuania (2):
  - Seamen' Hospital' Dept. of haematology, Klaipėda
  - Uni Hospital Santariskiu Clinic; Haematology, Vilnius
- Hospital Pulau Pinang, George Town, Pulau Pinang, Malaysia
- Mexico (4):
  - Instituto Biomedico De Investigacion A.C., Aguascalientes
  - Hospital Español; Hematología Sala 19, Mexico City
  - Col Instituto Tecnologico Y Estudios Superiores de Monterrey, Monterrey
  - Hospital Universitario Dr. Jose E. Gonzalez; Haematology, Monterrey
- New Zealand (3):
  - North Shore Hospital; Haematolgy, Auckland
  - Uni of Auckland; Dept of Molecular Medicine & Haematology, Auckland
  - Christchurch Hospital; Canterbury Health Laboratories, Christchurch
- Centro Hemato Oncologico Paitilla, Panama City, Panama
- Peru (5):
  - Hospital Nacional Almanzor Aguinaga Asenjo; Unidad De Investigacion Del Servicio De Oncologia Medica, Chiclayo
  - Hospital Nacional Edgardo Rebagliati Martins; Oncologia, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen; Oncology, Lima
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Hospital Nacional LNS dela Policia Nacional del Perú. Unidad Onco; Deapartamento de Oncología, Lima
- Philippines (3):
  - Cebu Cancer Institute; Perpetual Succour Hospital, Cebu
  - National Kidney and Transplant Institute; Chemotherapy Unit, Diliman, Quezon City
  - St Luke'S Medical Centre; Oncology, Quezon City
- Poland (8):
  - Szpital Specjalistyczny Podkarpacki Ośrodek Onkologiczny, Brzozów
  - Szpital Uniwersytecki W Krakowie; Klinika Hematologii, Krakow
  - Medical University School; Dept. of Haematology, Lodz
  - Katedra i Klinika Hematoonkologii i Transplantacji Szpiku; Uniwersytetu Medycznego w Lublinie, Lublin
  - Zaklad Opieki Zdrowotnej Mswia; Oddzial Chemioterapii, Olsztyn
  - Samodzielny Publiczny Centralny Szpital Kliniczny; Haematology Dept., Warsaw
  - Centralny Szpital Kliniczny Mswia; Klinika onkologii, hematologii i chorob wewnetrznych, Warsaw
  - Centrum Onkologii - Inst.Im. Marii Sklodowskiej-Curie; Lymphoma Dept., Warsaw
- Portugal (3):
  - HUC; Servico de Hematologia, Coimbra
  - IPO de Lisboa; Servico de Hematologia, Lisbon
  - Hospital de Sao Joao; Servico de Hematologia Clinica, Porto
- Russia (5):
  - Republican Clinical Oncologic Dispensary of Republic Of Tatarstan, Kazan'
  - N.N.Blokhin Russian Cancer Research Center; Dept. of Chemotherapy & Hemoblastosis, Moscow
  - Haematology Research Center; Haematology, Moscow
  - Semashko Central Clinical Hospital Moscow; Hematology, Moscow
  - Research Inst. of Hematology & Blood Transfusion ; Hematology, Saint Petersburg
- National Cancer Inst. ; Dept. of Chemotherapy, Bratislava, Slovakia
- South Korea (4):
  - Samsung Medical Centre; Oncology, Seoul
  - Asan Medical Center, Uni Ulsan Collegemedicine; Dept.Internal Medicine / Divisionhematology/Oncology, Seoul
  - Korean Cancer Center Hospital; Oncology, Seoul
  - Severance Hospital - Yonsei University; Medicine Dept., Seoul
- Spain (19):
  - Hospital Mutua de Terrassa; Servicio de Hematologia, Terrassa, Barcelona
  - Hospital Universitario Marques de Valdecilla; Servicio de Hematologia, Santander, Cantabria
  - Complejo Hospitalario Universitario A Coruña (CHUAC); Servicio de Hematologia, A Coruña, La Coruña
  - Hospital Universitario de Canarias;servicio de Oncologia, San Cristóbal de La Laguna, Tenerife
  - Hospital de Basurto; Servicio de Hematologia, Bilbao, Vizcaya
  - Hospital de Galdakano, Galdakano, Vizcaya
  - Hospital de la Santa Creu i Sant Pau; Servicio de Hematologia, Barcelona
  - Hospital Universitari Vall d'Hebron; Servicio de Hematologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital Duran i Reynals; Servicio de Hematologia, Barcelona
  - Complejo Hospitalario de Jaen- Hospital Universitario Medico Quirurgico; Servicio de Hematologia, Jaén
  - Hospital Universitario Clínico San Carlos; Servicio de Hematología, Madrid
  - Hospital Universitario la Paz; Servicio de Hematologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Hospital Clinico Universitario de Salamanca;Servicio de Hematologia, Salamanca
  - Hospital Universitario Virgen del Rocio; Servicio de Hematologia, Seville
  - Hospital Universitario la Fe; Servicio de Medicina Intena, Valencia
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
  - Hospital Universitario Miguel Servet; Servicio Hematologia, Zaragoza
- Sweden (4):
  - Skånes University Hospital, Skånes Department of Onclology, Lund
  - Skånes Universitetssjukhus; Kliniska Forskningsenheten Onkologimottagning medicinsk behandling, Malmo
  - Länssjukhuset; Medicinkliniken, Sundsvall
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- Universitätsspital Zürich; Klinik für Onkologie, Zurich, Switzerland
- Taiwan (3):
  - Veterans General Hospital; Division of Oncology, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center; Hemato-Oncology, Taipei
  - Chang Gung Medical Foundation-Taipei, Taoyuan District
- Thailand (6):
  - King Chulalongkorn Memorial Hospital; Division of Hematology, Department of Medicine, Bangkok
  - National Cancer Inst., Bangkok
  - Rajavithi Hospital; Medicine, Bangkok
  - Siriraj Hospital; Division of Hematology, Department of Medicine, Bangkok
  - Chiang Mai Uni Hospital; Division of Hematology,Dept of Medicine,Faculty of Medicine, Chiang Mai
  - Srinagarind Hospital, Khon Kaen Uni ; Dept of Medicine, Khon Kaen
- United Kingdom (12):
  - Birmingham Heartlands Hospital; Department of Haematology, Birmingham
  - Bradford Royal Infirmary; Haematology Department, Bradford
  - North Hampshire Hospital; Dept. of Haematology, Hampshire
  - Princess Alexandra Hospital; Department of Haematology, Harlow
  - Leicester Royal Infirmary; Dept. of Medical Oncology, Leicester
  - Royal Liverpool Uni Hospital; Haematology, Liverpool
  - St. George'S Hospital; Haematology, London
  - Hillingdon Hospital, Middx
  - Churchill Hospital; Oxford Cancer and Haematology Centre, Oxford
  - Royal Hallamshire Hospital; Haematology Dept, Sheffield
  - Weston Park Hospital; Cancer Clinical Trials Centre, Sheffield
  - The Royal Wolverhampton Hospitals NHS Trust; Department of Haematology, Wolverhampton

REFERENCES:
- [Derived] McCord R, Bolen CR, Koeppen H, Kadel EE 3rd, Oestergaard MZ, Nielsen T, Sehn LH, Venstrom JM. PD-L1 and tumor-associated macrophages in de novo DLBCL. Blood Adv. 2019 Feb 26;3(4):531-540. doi: 10.1182/bloodadvances.2018020602. PMID 30770362
- [Derived] Seymour JF, Pfreundschuh M, Trneny M, Sehn LH, Catalano J, Csinady E, Moore N, Coiffier B; MAIN Study Investigators. R-CHOP with or without bevacizumab in patients with previously untreated diffuse large B-cell lymphoma: final MAIN study outcomes. Haematologica. 2014 Aug;99(8):1343-9. doi: 10.3324/haematol.2013.100818. Epub 2014 Jun 3. PMID 24895339

RESULTS

PARTICIPANT FLOW:
Period: Treatment
Arm/Group | Bevacizumab + Rituximab + CHOP | Placebo + Rituximab + CHOP
Started | 390 | 397
Completed | 203 | 260
Not Completed | 187 | 137
Not completed — Adverse event/intercurrent illness | 86 | 39
Not completed — Insufficient therapeutic response | 37 | 39
Not completed — Death | 17 | 10
Not completed — Withdrew consent | 15 | 12
Not completed — Administrative/reason not specified | 17 | 21
Not completed — Refused treatment | 10 | 7
Not completed — Violation of selection criteria at entry | 3 | 3
Not completed — Other protocol violation | 1 | 5
Not completed — Failure to return | 1 | 1
Period: Safety Follow-up
Arm/Group | Bevacizumab + Rituximab + CHOP | Placebo + Rituximab + CHOP
Started | 203 | 260
Completed | 64 | 142
Not Completed | 139 | 118
Not completed — Insufficient therapeutic response | 40 | 50
Not completed — Death | 40 | 29
Not completed — Withdrew consent | 32 | 23
Not completed — Failure to return | 9 | 6
Not completed — Administrative/not specified | 8 | 6
Not completed — Refused treatment/did not cooperate | 6 | 4
Not completed — Adverse event/intercurrent illness | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + Rituximab + CHOP | Placebo + Rituximab + CHOP | Total
Number analyzed (Participants) | 390 | 397 | 787
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.89 (14.256) | 56.98 (15.399) | 57.44 (14.841)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 193 | 400
  Male | 183 | 204 | 387

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of disease progression (PD)/relapse, as determined by the investigator, or death from any cause, whichever occurred earlier. A patient with PD/relapse must meet at least 1 of the following criteria: (1) Appearance of any new lesion > 1.0 cm in the short axis during or at the end of therapy. (2) ≥ 50 % increase from nadir in the sum of the products of diameters (SPD, maximum diameter of a tumor x largest diameter perpendicular to the maximum diameter) of any previously involved nodes, in a single involved node, or the size of other lesions (eg, splenic or hepatic nodules). To be considered progressive disease, a lymph node with a diameter of the short axis < 1.0 cm must increase by ≥ 50% to a size of 1.5 x 1.5 cm or > 1.5 cm in the long axis. (3) ≥ 50 % increase in the greatest diameter of any previously identified node > 1.0 cm in its short axis or in the SPD of more than 1 node.
Time Frame: Baseline to end of the study (up to 4 years, 4 months)
Population: Intent-to-treat population: All randomized patients, regardless whether or not they had actually received the assigned treatments.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Bevacizumab + Rituximab + CHOP | Placebo + Rituximab + CHOP
Number analyzed (Participants) | 390 | 397
Months | 40.2 [12.1 to NA] — The 75th percentile could not be estimated due to a lack of events. | 42.9 [13.6 to NA] — The 75th percentile could not be estimated due to a lack of events.

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of death due to any cause.
Time Frame: Baseline to end of the study (up to 4 years, 4 months)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Bevacizumab + Rituximab + CHOP | Placebo + Rituximab + CHOP
Number analyzed (Participants) | 390 | 397
Months | NA [34.0 to NA] — The median and 75th percentile could not be estimated due to a lack of events, | NA [42.9 to NA] — The median and 75th percentile could not be estimated due to a lack of events,

3. Secondary Outcome: Overall Response (OR) Assessed According to the Revised Response Criteria for Malignant Lymphoma
Description: OR = a complete response (CR), an unconfirmed CR, or a partial response (PR). CR = Complete disappearance of disease and disease-related symptoms. All lymph nodes and nodal masses regressed on computed tomography (CT) to normal size (≤ 1.5 cm in their greatest transverse diameter for nodes > 1.5 cm prior to therapy and ≤ 1.0 cm in their short axis for nodes 1.1-1.5 cm in their long axis and > 1.0 cm in their short axis prior to therapy). Spleen and/or liver not palpable on physical examination, normal size by imaging, and disappearance of nodules related to lymphoma. If bone marrow was involved prior to therapy, infiltrate must have cleared on repeat biopsy. PR = ≥ 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses. No increase in the size of the other nodes, liver, or spleen. Splenic and hepatic nodules regressed by ≥ 50% in their SPD or, for single nodules, in the greatest transverse diameter. No new sites of disease.
Time Frame: At the end of treatment (Cycle 8, up to 12 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Bevacizumab + Rituximab + CHOP | Placebo + Rituximab + CHOP
Number analyzed (Participants) | 390 | 397
Percentage of patients | 63.1 | 70.5

ADVERSE EVENTS:
Time Frame: All adverse events (AE) were reported starting from the first dose up to 92 days after the last dose of study drug. AEs of special interest were reported up to 6 months after the last dose.
Description: Safety analysis population: All patients who received at least 1 dose of study drug whether withdrawn prematurely or not. Bevacizumab (B) 395=390 randomized-2 no treatment+7 randomized to placebo who received B. Placebo to B 386=397 randomized-5 no treatment-7 received B+1 randomized to B who received placebo but no B.
Arm/Group | Bevacizumab + Rituximab + CHOP | Placebo + Rituximab + CHOP
Serious Adverse Events (participants affected / at risk) | 224/395 | 173/386
Other Adverse Events (participants affected / at risk) | 346/395 | 331/386
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Rituximab + CHOP (N=395) | Placebo + Rituximab + CHOP (N=386)
Febrile neutorpenia (Blood and lymphatic system disorders) | 63 | 48
Neutropenia (Blood and lymphatic system disorders) | 12 | 17
Leukopenia (Blood and lymphatic system disorders) | 6 | 5
Anaemia (Blood and lymphatic system disorders) | 8 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 4
Agranulocytosis (Blood and lymphatic system disorders) | 3 | 2
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 3
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 22 | 16
Septic shock (Infections and infestations) | 6 | 4
Infection (Infections and infestations) | 3 | 6
Urinary tract infection (Infections and infestations) | 6 | 3
Bronchopneumonia (Infections and infestations) | 2 | 6
Gastroenteritis (Infections and infestations) | 2 | 4
Neutropenic sepsis (Infections and infestations) | 5 | 1
Sepsis (Infections and infestations) | 2 | 4
Neutropenic infection (Infections and infestations) | 1 | 4
Device related infection (Infections and infestations) | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Anal abscess (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 0 | 2
Escherichia sepsis (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 1 | 1
Oesophageal candidiasis (Infections and infestations) | 2 | 0
Pharyngitis (Infections and infestations) | 1 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 2 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0
Amoebiasis (Infections and infestations) | 1 | 0
Appendiceal abscess (Infections and infestations) | 0 | 1
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 1
Fungal oesophagitis (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Gastrointestinal fungal infection (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 1
Infectious peritonitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Lymph gland infection (Infections and infestations) | 1 | 0
Lymphadenitis bacterial (Infections and infestations) | 0 | 1
Meningitis cryptococcal (Infections and infestations) | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Oral infection (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0
Pneumocystis jiroveci infection (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Splenic abscess (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Systemic candida (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tuberculous pleurisy (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 15 | 5
Cardiac failure (Cardiac disorders) | 6 | 4
Cardiac failure congestive (Cardiac disorders) | 5 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 4
Angina pectoris (Cardiac disorders) | 1 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiotoxicity (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Ventricular hypokinesia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 3
Ascites (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 2 | 2
Gastric perforation (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Periodontitis (Gastrointestinal disorders) | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 14 | 15
Asthenia (General disorders) | 4 | 2
Chest pain (General disorders) | 0 | 3
Death (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 3 | 0
Fatigue (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 2 | 0
Catheter site haemorrhage (General disorders) | 1 | 0
Effusion (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Medical device complication (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 3
Syncope (Nervous system disorders) | 0 | 4
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Convulsion (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Hypertension (Vascular disorders) | 6 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 4
Hypertensive crisis (Vascular disorders) | 2 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Chemical injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Ejection fraction decreased (Investigations) | 4 | 3
C-reactive protein increased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Multiple gated acquisition scan abnormal (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 2
Anaphylactic reaction (Immune system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Aplasia (Congenital, familial and genetic disorders) | 1 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Rituximab + CHOP (N=395) | Placebo + Rituximab + CHOP (N=386)
Nausea (Gastrointestinal disorders) | 107 | 106
Diarrhoea (Gastrointestinal disorders) | 95 | 81
Constipation (Gastrointestinal disorders) | 88 | 70
Vomiting (Gastrointestinal disorders) | 56 | 70
Stomatitis (Gastrointestinal disorders) | 33 | 36
Dyspepsia (Gastrointestinal disorders) | 23 | 35
Abdominal pain (Gastrointestinal disorders) | 32 | 25
Abdominal pain upper (Gastrointestinal disorders) | 17 | 32
Haemorrhoids (Gastrointestinal disorders) | 23 | 12
Fatigue (General disorders) | 71 | 71
Pyrexia (General disorders) | 71 | 55
Asthenia (General disorders) | 59 | 60
Mucosal inflammation (General disorders) | 61 | 45
Oedema peripheral (General disorders) | 24 | 29
Neutropenia (Blood and lymphatic system disorders) | 88 | 119
Anaemia (Blood and lymphatic system disorders) | 66 | 96
Leukopenia (Blood and lymphatic system disorders) | 42 | 49
Thrombocytopenia (Blood and lymphatic system disorders) | 24 | 30
Headache (Nervous system disorders) | 59 | 59
Neuropathy peripheral (Nervous system disorders) | 38 | 38
Paraesthesia (Nervous system disorders) | 42 | 31
Peripheral sensory neuropathy (Nervous system disorders) | 25 | 28
Dizziness (Nervous system disorders) | 24 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 43
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 47 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 27
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 27 | 19
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 24 | 14
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 29 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 96 | 80
Rash (Skin and subcutaneous tissue disorders) | 22 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 37
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 19
Bone pain (Musculoskeletal and connective tissue disorders) | 23 | 17
Nasopharyngitis (Infections and infestations) | 30 | 22
Urinary tract infection (Infections and infestations) | 24 | 23
Upper respiratory tract infection (Infections and infestations) | 25 | 17
Decreased appetite (Metabolism and nutrition disorders) | 60 | 46
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 17
Hypertension (Vascular disorders) | 54 | 12
Insomnia (Psychiatric disorders) | 29 | 30
Weight decreased (Investigations) | 24 | 21

LIMITATIONS AND CAVEATS:
Due to premature termination of the study, the efficacy results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.